CLINICAL TRIAL: NCT06398002
Title: The Effect of Increasing Dialysate Calcium on Serum Calcification Propensity in Subjects With Secondary Hyperparathyroidism and End-Stage Kidney Disease
Brief Title: The Effect of Increasing Dialysate Calcium on T50 in Subjects With Secondary Hyperparathyroidism and ESKD
Acronym: CaT50HD
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Iain Bressendorff (Other)
Responsible Party: Sponsor-Investigator, Iain Bressendorff, MD PhD, Herlev Hospital
Organization: Herlev Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CaT50HD
Record Dates: First submitted 2024-04-30; First posted 2024-05-03 (Actual); Last update posted 2024-05-03 (Actual); Status verified 2024-04

CONDITIONS: Secondary Hyperparathyroidism; End-stage Kidney Disease
MeSH Terms: conditions — Hyperparathyroidism, Secondary; Kidney Failure, Chronic

STUDY DESIGN:
Intervention Model Description: Randomised, double-blind, parallel-group, controlled clinical trial
Who Masked: Participant, Investigator
Masking Description: Blinding of participants and investigators. Dialysis nurses will be aware of treatment assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dialysate calcium 1.25 mmol/L (standard) (Active Comparator)
  Interventions: Other: Dialysate calcium 1.50 mmol/L
- Dialysate calcium 1.50 mmol/L (high) (Experimental)
  Interventions: Other: Dialysate calcium 1.50 mmol/L

INTERVENTIONS:
Other: Dialysate calcium 1.50 mmol/L — Increased dialysate calcium of 1.50 mmol/L (as compared to standard dialysate calcium of 1.25 mmol/L)

SUMMARY:
Patients with end-stage kidney disease (ESKD) have an increased risk of cardiovascular mortality. High parathyroid hormone (PTH) from secondary hyperparathyroidism leads to increased efflux of phosphate and calcium from bone, which exacerbates vascular calcification and increases the risk of bone fractures. The main driving factor for secondary hyperparathyroidism is hypocalcaemia caused by low levels of 1,25-dihydroxy vitamin D and pharmacological supplementation with activated vitamin D and oral calcium-containing phosphate-binders are used to control secondary hyperparathyroidism. The amount of calcium used in this context is controversial, as higher calcium load in blood may theoretically increase vascular calcification. Conversely, by alleviating the efflux of phosphate and calcium from bone due to secondary hyperparathyroidism, increasing the load of calcium might actually prevent vascular calcification.

To study this further, we wish to conduct a randomised double-blinded controlled clinical trial of increasing dialysate Ca from 1.25 mmol/L (standard dialysate concentration) to 1.50 mmol/L in patients with ESKD and secondary hyperparathyroidism on maintenance haemodialysis (HD). The overall effect of increased dialysate calcium will be gauged by its effect on serum calcification propensity (T50) and on markers of bone turnover.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Treatment with thrice-weekly maintenance HD for ESKD for > 3 months.
* Dialysate calcium of 1.25 mmol/L (standard concentration).
* Plasma ionised calcium < 1.35 mmol/L (average of last 3 months).
* Plasma intact PTH > 14 ρmol/L.
* Plasma total alkaline phosphatase >90 U/L
* Negative pregnancy test and use of highly effective and safe contraception.
* Able to give written informed consent.

Exclusion Criteria:

* Treatment with peritoneal dialysis.
* Clinical bone fracture within the last 6 months.
* Treatment with bisphosphonates, denosumab, romosozumab, or teriparatide within the last 3 months.
* Other diseases or conditions, which, in the opinion of the site investigator, would prevent participation in or completion of the trial.
* Pregnancy or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2024-08-01 (Estimated); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Difference in serum calcification propensity (T50) | 28 days
  Between-groups difference in T50 at day 28 adjusted for T50 at day 0

SECONDARY OUTCOMES:
Difference in bone-specific alkaline phosphatase (bALP) | 28 days
  Between-groups difference in bALP at day 28 adjusted for bALP at day 0
Difference in procollagen 1 intact N-terminal propeptide (P1NP) | 28 days
  Between-groups difference in P1NP at day 28 adjusted for P1NP at day 0
Difference in tartrate-resistant acid phosphatase 5b (TRAcP 5b) | 28 days
  Between-groups difference in TRAcP 5b at day 28 adjusted for TRAcP 5b at day 0
Difference in parathyroid hormone (PTH) | 28 days
  Between-groups difference in PTH at day 28 adjusted for PTH at day 0
Difference in calciprotein monomers (CPM) | 28 days
  Between-groups difference in CPM at day 28 adjusted for CPM at day 0
Difference in primary calciprotein particles (CPP-1) | 28 days
  Between-groups difference in CPP-1 at day 28 adjusted for CPP-1 at day 0
Difference in primary calciprotein particles (CPP-2) | 28 days
  Between-groups difference in CPP-2 at day 28 adjusted for CPP-2 at day 0
Difference in plasma ionised calcium (iCa) | 28 days
  Between-groups difference in iCa at day 28 adjusted for iCa at day 0
Difference in plasma phosphate (PO4) | 28 days
  Between-groups difference in PO4 at day 28 adjusted for PO4 at day 0
Difference in plasma magnesium (Mg) | 28 days
  Between-groups difference in Mg at day 28 adjusted for Mg at day 0
Difference in all above variables | 28 days
  Within-groups difference in all above variables at day 28 adjusted for values at day 0

CONTACTS AND LOCATIONS:
Overall Officials: Iain Bressendorff, MD PhD, Principal Investigator — Herlev and Gentofte Hospital

IPD SHARING:
Plan to Share IPD: Yes
Upon reasonable request to the investigators
Supporting Information: Study Protocol, SAP